CLINICAL TRIAL: NCT04575987
Title: How Bariatric Surgery Impacts Pelvic Floor Disorders Evolution : Analysis on a Cohort From a French Hospital.
Brief Title: Long Term Effect of Bariatric Surgery on Pelvic Floor Disorders
Acronym: ICONES
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-A02219-30
Record Dates: First submitted 2020-09-16; First posted 2020-10-05 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Bariatric Surgery Candidate; Weight Loss
MeSH Terms: conditions — Weight Loss | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire — Questionnaires will be sent by email or by post, in which questions about PFD, obstetrical history or dietetic follow-up will be asked.
  Some obstetrical issues will be get from women medical files.

SUMMARY:
Bariatric surgery is increasingly practiced, as it is the most efficient treatment for morbid obesity. More than eighty percent of the operated patients are women. Nethertheless, few is known about gynecologic long-term impact of such surgeries, especially regarding pelvic floor disorders (PFD). This work aims at studying the evolution of PFD in women following a bariatric surgery more than 18 months ago in a French university center Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Women,
* aged from 18 to 50 years old the day of their surgery,
* had a bariatric surgery in Poitiers university hospital center (France),
* are under french social security system.

Exclusion Criteria:

* to be under guardianship or tutelage measures
* to express opposition to participate to this study.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women had a bariatric surgery in Poitiers university hospital center (France)
Sampling Method: Non-Probability Sample
Enrollment: 709 (Estimated)
Dates: Start 2020-12-14 (Actual); Primary Completion 2021-06-14 (Estimated); Study Completion 2021-06-14 (Estimated)

PRIMARY OUTCOMES:
Prevalence of the main PFD | minimum 18 months after surgery
  To evaluate the prevalence of the main PFD regarding the efficiency of the bariatric surgery 18 months or more after. The prevalence of PFD will be estimated thanks to the PFDI-20 questionnaire :
  * urinary incontinence : at least one positive answer to questions 16 to 18 of PFDI-20
  * bowel incontinence : at least one positive answer to questions 8 to 10 of PFDI-20
  * vaginal prolapse : positive answer to question 3 of PFDI-20 Efficiency of the bariatric surgery will be estimated thanks to the weight registered in the medical file before bariatric surgery and the most recent weight obtained thanks to the questionnaire.
  Our results will be adjusted for age, menopausal status, obstetrical and surgical history.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Poitiers, Poitiers, France